CLINICAL TRIAL: NCT05442476
Title: Effects of Kinesio-Taping and Muscle Energy Technique on Chronic Sacroiliac Joint Dysfunction Among Postpartum Females- A Randomized Controlled Trial
Brief Title: Effects of Kinesio-Taping and Muscle Energy Technique on Chronic Sacroiliac Joint Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziauddin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5490522REH
Record Dates: First submitted 2022-06-22; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Musculoskeletal Injury
Keywords: Sacroiliac joint; Exercise; Muscle energy technique
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotaping (Experimental)
  Interventions: Other: Kinesiotaping; Other: conventional physiotherapy
- Muscle Energy Technique (Other)
  Interventions: Other: Muscle Energy Technique; Other: conventional physiotherapy

INTERVENTIONS:
Other: Kinesiotaping — For the KT application, participants will be asked to stand with keeping their feet at shoulder level in a comfortable manner. The patient will be in a standing position with lumbar spine flexion. A 5 cm wide long I-shaped piece of tape will be applied with 80% tension transverse to the patient's painful area and the bilateral SIJ region, with no tension applied to the ends of the tape. Another short piece of tape will be applied with 80% tension at an angle from the painful point to the hip, and no tension will be applied to the ends of the tape. An identical application will be performed on the other side of the sacroiliac region
  Arms: kinesiotaping
Other: Muscle Energy Technique — The subject will be asked for the sitting on the treatment table, back towards the therapist. Then the subject will be taken into flexion, rotation and side bending. When the subject will reach the tolerated limit of flexion, the therapist will ask him to perform extension, sidebending and rotation to the opposite side while holding the breath for 7-10 seconds and rest for 2-3 seconds, then the patient will be asked to release the breath. The therapist will wait for the participant's full exhalation and then will take her further in all the directions of restriction, towards the new barrier. MET will be performed for 10 repetitions.
  Arms: Muscle Energy Technique
Other: conventional physiotherapy — conventional physiotherapy

SUMMARY:
Pregnancy is the main occasion of every woman's life in which numerous episodes of physiological and anatomical adjustments takes place within woman's body to become a mother. Anatomical changes often leads to poor biomechanics and may cause mechanical dysfunction of spine especially lower back.. Sacroiliac joint (SIJ) goes through most of mobility during the period of pregnancy due to hormone release causes ligamentous laxity that can cause SIJD.

DETAILED DESCRIPTION:
Fifty two patients will be randomly divided into two groups i.e. Group-A (n=26) and B (n=26) respectively through simple random sampling, sealed envelope method. Informed consent will be taken from the participant prior to intervention. Baseline assessment will be carried out before the first session of all the recruited participants on four outcome measures using, Patrick's FABER test for provocation of pain, NPRS for intensity of pain, RMDQ for physical disability and PALM Pelvic Inclinometer for pelvic asymmetry respectively. Skin reaction test will be conducted before randomization after the baseline assessment for all participants. A small patch of kinesio tape will be applied to the hip region and the participants will be asked to keep it for 24 hours. If any of the participants will develop allergic reaction, it will be removed immediately and participants with positive results will be excluded from the study. After this test, the allergy-free patients will be randomized into 2 groups for treatment. Participants of Group-A will be applied KT with conventional physiotherapy while Group-B participants will perform MET with conventional physiotherapy. Whereas, both the groups will be given 12 sessions of their respective protocol, comprising 20 minutes, 3 times/week for the duration of 4 weeks. After the end of the intervention, subjects will be reassessed after the last session and data will be collected on the same outcome measures for further evaluation

ELIGIBILITY:
Inclusion Criteria:

* Postpartum with diagnosed cases of SIJD dysfunction (after 3 months of delivery) with age range between 20 to 35 years
* Postpartum with unilateral/bilateral both SIJD
* Postpartum with anterior innominate

Exclusion criteria:

* History of any fracture at lower limb in recent 6 months
* Pregnant females
* Spinal stenosis, spondylolisthesis
* Malignancy of spine or lower limb
* Radiculopathy
* Conditions like diastasis recti, prolapse pelvic organ
* History of recent infection

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2022-06-18 (Actual); Primary Completion 2022-09-24 (Estimated); Study Completion 2022-10-10 (Estimated)

PRIMARY OUTCOMES:
Disability | Baseline
  It will be used for the participants to assess the disability with low back pain, comprised of 24 items regarding functional status that are likely to be affected by LBP. The scoring of RMQD will show '0' as no disability and '24' as maximum disability
Disability | After 4 weeks
  It will be used for the participants to assess the disability with low back pain, comprised of 24 items regarding functional status that are likely to be affected by LBP. The scoring of RMQD will show '0' as no disability and '24' as maximum disability
Pelvic tilting | Baseline
  PALM device is portable, convenient to use that combines the features of a caliper and inclinometer. It is reliable tool used for measuring pelvic tilting angle/inclination by marking a point just inferior to ASIS; another mark inferior to PSIS. Keeping the calipers of the PALM on these two points to determine the distance in centimeter between two points
Pelvic tilting | After 4 weeks
  PALM device is portable, convenient to use that combines the features of a caliper and inclinometer. It is reliable tool used for measuring pelvic tilting angle/inclination by marking a point just inferior to ASIS; another mark inferior to PSIS. Keeping the calipers of the PALM on these two points to determine the distance in centimeter between two points

CONTACTS AND LOCATIONS:
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan